CLINICAL TRIAL: NCT05623150
Title: CHronic Hepatopathies Associated with ALcohol Consumption and MetAbolic Syndrome
Acronym: CHALNA2
Status: Recruiting | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: C20-12
Record Dates: First submitted 2021-12-27; First posted 2022-11-21 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-02

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Non-Alcoholic Steatohepatitis; Alcohol-related Liver Disease; Cirrhosis, Liver; Hepatocellular Carcinoma
Keywords: Non-Alcoholic Fatty Liver Disease; Non-Alcoholic Steatohepatitis; Alcohol-related Liver Disease; Cirrhosis, Liver; Hepatocellular Carcinoma
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Cirrhosis; Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — standard liver biopsy (for immunocytochemistry), frozen liver biopsy, frozen serum, frozen plasma, DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Descriptive study: The patients included in this observational study are patients with hepatic steatosis either related to NAFLD or to alcohol-related liver disease.
  Patients included in the study may have hepatocellular carcinoma.
  Thus, 4 groups of patients can be recruited:
  * patients with NAFLD without hepatocellular carcinoma,
  * patients with NAFLD with hepatocellular carcinoma,
  * patients with alcohol-related liver disease without hepatocellular carcinoma, -patients with alcohol-related liver disease with hepatocellular carcinoma.
  Interventions: Diagnostic Test: Liver biopsy

INTERVENTIONS:
Diagnostic Test: Liver biopsy — Liver biopsy planned as part of routine care. Clinical-biological characterisation with bio collections.

SUMMARY:
The aim is to determine the metabolic factors, host immune factors, and medical imaging data associated with the development of HepatoCellular Carcinoma (HCC) in patients with alcohol-related liver disease or dysmetabolic steatosis/Non-Alcoholic SteatoHepatitis.

The investigators will include patients with and without cirrhosis in order to identify early molecular mechanisms involved in the development of HCC especially in non-cirrhotic patients.

DETAILED DESCRIPTION:
Type and methodology of the research:

Within the framework of the usual management of the patient's pathology, a clinico-biological characterization (dietary and physical activity questionnaires, "performans status", anthropometric measurements, usual blood biology characterizing the hepatic, renal and inflammatory function, the carbohydrate and lipid metabolism, the non invasive test for liver fibrosis ELF etc.) will be carry out. In order to collect radiomic data, liver imaging (particularly in case of HCC) will be done.

A liver biopsy and constitution of a biobank (samples of plasma, sera, DNA and leucocyte pellets) will be performed.

The elements necessary for the classification of possible hepatocellular carcinomas (BCLC classification) will be collected.

Anticipated research schedule:

* The duration of inclusion in this research will be 10 years.
* The duration of the patient's participation will be from 1 day (if the consent is signed and the biopsy is performed on the same day) to 2 months (maximum reflection period is 8 weeks between the signature of the consent and the taking of samples).
* The total duration of the research (from the first inclusion, to the last visit of the last participant) will be 10 years and 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Criteria common to all patients:

  1. Affiliation to French social security.
  2. Male or female ≥ 18 years of age
  3. Patients able to receive and understand information about the research and to give written informed consent duly signed by the patient and the investigator (at the latest on the day of inclusion and before any examination necessary for the research).
* Patients in the NAFLD group with HCC:

  1. Alcohol consumption ≤ 30 g pure alcohol/d (or 210 g pure alcohol/week) for men and ≤ 20 g pure alcohol/d (140 g pure alcohol/week) for women.
  2. Decision, less than 3 months old, of liver biopsy of the suspected HCC nodule and non-tumour liver tissue performed as a clinical routine.
  3. No systemic treatment for HCC within 6 months prior to inclusion.
* Patients in the NAFLD group without HCC:

  1. Alcohol consumption ≤ 30 g pure alcohol/d (or 210 g pure alcohol/week) for men and ≤ 20 g pure alcohol/d (140 g pure alcohol/week) for women.
  2. Decision of less than 3 months of a liver biopsy performed as a clinical routine. Biopsy will be motivated by liver function disturbance(s) and/or ultrasound steatosis given the lack of validated non-invasive tests or the lack of accuracy (grey areas) of available non-invasive tests for the diagnosis of necro-inflammation and/or fibrosis in some of these patients.
* Patients in the alcohol-related liver disease group with HCC:

  1. Alcohol consumption > 30 g pure alcohol/d (or 210 g pure alcohol/week) for men and > 20 g pure alcohol/d (140 g pure alcohol/week) or binge drinking
  2. Decision within 3 months of liver biopsy of suspected HCC nodule and non-tumour liver tissue performed as part of clinical routine
  3. No systemic treatment for HCC within 6 months prior to inclusion.
* Patients in the alcohol-related liver disease group without HCC:

  1. Alcohol consumption > 30 g pure alcohol/d (or 210 g pure alcohol/week) for men and > 20 g pure alcohol/d (140 g pure alcohol/week) or binge drinking
  2. Decision of less than 3 months for a liver biopsy to be performed as a clinical routine. Biopsy will be motivated by liver balance disturbance(s) and/or ultrasound steatosis given the lack of validated non-invasive tests or the lack of accuracy (grey areas) of available non-invasive tests for the diagnosis of necro-inflammation and/or fibrosis in some of these patients.

Exclusion Criteria:

1. Positive HIV serology
2. Patients with detectable hepatitis C viral load
3. Presence of Hbs antigen
4. History of autoimmune hepatitis type 1 or 2, primary biliary cholangitis, primary sclerosing cholangitis, Wilson's disease, genetic haemochromatosis homozygous, alpha1 anti-trypsin deficiency
5. Long-term use of methotrexate, corticosteroids, anti-Tumor Necrosis Factor cyclosporine, tacrolimus
6. History of solid organ transplantation or bone marrow transplantation
7. Cancerous disease in the process of being treated, except for skin cancer (excluding melanoma)
8. Patients under legal protection or unable to express their consent,
9. Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients included in this observational study are patients with hepatic steatosis either related to NAFLD or to alcohol-related liver disease.
  Patients included in the study may have hepatocellular carcinoma. Thus, 4 groups of patients can be recruited: patients with NAFLD without hepatocellular carcinoma, patients with NAFLD with hepatocellular carcinoma, patients with alcohol-related liver disease without hepatocellular carcinoma, patients with alcohol-related liver disease with hepatocellular carcinoma.
Sampling Method: Non-Probability Sample
Enrollment: 710 (Estimated)
Dates: Start 2022-12-06 (Actual); Primary Completion 2032-01 (Estimated); Study Completion 2032-03 (Estimated)

PRIMARY OUTCOMES:
Primary outcome measure CHALNA2 | 2022-2032
  The primary endpoint will be the study of variations in metabolic gene markers (i.e. mRNA of genes implicated in inflammation or metabolism assessed in qPCR, using a housekeeping gene such as glyceraldehyde-3-phosphate dehydrogenase (GAPDH)), in patients with and without hepatocellular carcinoma with different levels of severity of liver damage.

SECONDARY OUTCOMES:
Secondary outcome measure CHALNA2 | 2022-2032
  Secondary endpoint will include variations in other gene markers (e.g. genes implicated in the regeneration, cell deaths and tumor, assessed in qPCR, using a housekeeping gene such as glyceraldehyde-3-phosphate dehydrogenase (GAPDH)) in patients with and without hepatocellular carcinoma with different levels of severity of liver damage.
3th outcome measure CHALNA2 | 2022-2032
  3th endpoint will include variations in genetic markers (Single Nucleotide Polymorphisms (SNPs)), in patients with and without hepatocellular carcinoma with different levels of severity of liver damage.
  The frequency of SNPs will be compared to that found in the UK biobank cohort.
4th outcome measure CHALNA2 | 2022-2032
  4th endpoint will include variations in epigenetic markers (histone methylation, micro RNA), in patients with and without hepatocellular carcinoma with different levels of severity of liver damage.
5th outcome measure CHALNA2 | 2022-2032
  5th endpoint will include variations in tissue proteins (including tumor and non tumor tissue), in patients with and without hepatocellular carcinoma with different levels of severity of liver damage. Western blots will be quantified and compared in an automated way.
6th outcome measure CHALNA2 | 2022-2032
  6th endpoint will include variations in specific markers or markers derived from analysis via platforms (OMICS), in patients with and without hepatocellular carcinoma with different levels of severity of liver damage.
7th outcome measure CHALNA2 | 2022-2032
  7th endpoint will include variations in radiomics (radiomics is a method that extracts a large number of features from medical images using data-characterisation algorithms), in patients with and without hepatocellular carcinoma with different levels of severity of liver damage.

CONTACTS AND LOCATIONS:
Locations (1):
- Batiment Archimed 151, route de Saint Antoine de Ginestière, Nice, France

IPD SHARING:
Plan to Share IPD: No